CLINICAL TRIAL: NCT00990080
Title: Safety and Immunogenicity of Two Mixed Primary Immunization Schedules: Pediacel® at 2 and 4 Months of Age Followed by One Dose of Infanrix™ IPV/Hib at 6 Months of Age; and, Infanrix™ IPV/Hib at 2 Months of Age, Followed by Pediacel® at 4 and 6 Months of Age
Brief Title: Interchangeability of Infanrix™ IPV/Hib and Pediacel® at 2,4 & 6 Months of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dalhousie University (Other)
Collaborators: IWK Health Centre (Other); MCM Vaccines B.V. (Industry)
Responsible Party: Dr Joanne Langley, Canadian Center for Vaccinology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SP91
Record Dates: First submitted 2009-10-05; First posted 2009-10-06 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2011-06

CONDITIONS: Infant Immunizations
MeSH Terms: interventions — diphtheria-tetanus-five component acellular pertussis-inactivated poliomyelitis -Haemophilus influenzae type b conjugate vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): Pediacel® at 2 and 4 months of age followed by Infanrix™-IPV/Hib at 6 months.
  Interventions: Biological: Pediacel® and Infanrix™-IPV/Hib
- Group 2 (Active Comparator): Infanrix™-IPV/Hib at 2 months of age followed by Pediacel® at 4 and 6 months.
  Interventions: Biological: Pediacel® and Infanrix™-IPV/Hib

INTERVENTIONS:
Biological: Pediacel® and Infanrix™-IPV/Hib — 0.5 mL IM at 2,4 and 6 months of age

SUMMARY:
To demonstrate the safety and immunogenicity of two mixed primary immunization schedules: Pediacel® at 2 and 4 months of age followed by one dose of Infanrix™ IPV/Hib at 6 months of age; and, Infanrix™ IPV/Hib at 2 months of age, followed by Pediacel® at 4 and 6 months of age.

DETAILED DESCRIPTION:
Immunogenicity will be evaluated using the following:

Serological outcome measures will be assessed on day 0 (visit 1) and 28-42 days after the 3rd dose of the primary series for both groups:

* Seroprotection rates for antibodies against PRP (anti-PRP), defined as percentage of subjects with antibody concentrations ≥ 0.15 µg/ml and ≥ 1.0 µg/ml.
* Geometric mean concentration (GMC) for antibodies against PT, FHA, PRN, and FIM.
* Anti-pertussis antibody concentrations ≥4-fold rise (post-Dose 3/pre-Dose 1).

Safety will be evaluated using the following:

* Occurrence, time to onset, number of days of occurrence, severity and seriousness of solicited injection site reactions (tenderness, erythema, swelling) and systemic symptoms (fever, vomiting, crying abnormal, drowsiness, appetite decreased, irritability) within 8 days (Day 0 - Day 7) after each vaccination and across all vaccinations.
* Occurrence, nature, time to onset, duration, severity, and relationship to vaccination of unsolicited adverse events (AE) occurring within 31 days (Day 0 -Day 30) of each vaccination.
* Occurrence, nature, time to onset, duration, and relationship to vaccination of any serious adverse events (SAE) during the entire study period for all groups.

ELIGIBILITY:
Inclusion Criteria:

1. Infants aged 6 wks (42 days) to 2 months (1 day before they turn 3 months) inclusive on the day of inclusion.
2. Born at full term of pregnancy (defined as ≥37 weeks, 0 days).
3. Informed consent form signed by the parent(s) or legally authorized representative.
4. Able to attend all scheduled visits and to comply with the study procedures.
5. Parent or legally authorized representative has access to a telephone.
6. Parent or legally authorized representative able to read and write in English or French.

Exclusion Criteria:

1. Participation in another clinical trial in the 4 weeks preceding the first trial vaccination.
2. Planned participation in another clinical trial during the present trial period.
3. Personal history of congenital or acquired immunodeficiency, immunosuppressive therapy such as long-term systemic corticosteroids therapy.
4. Known or suspected systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to a vaccine containing the same substances as the trial vaccine(s).
5. Chronic illness that could interfere with trial conduct or completion.
6. Received blood or blood-derived products since birth.
7. Any vaccination preceding the first trial vaccination, except vaccinations recommended as part of the infant schedule.
8. Previous vaccination with any acellular pertussis- (DTaP) or whole cell pertussis-DTwP) based combination vaccines, Haemophilus influenzae type b Hib)conjugate,or poliovirus vaccines.
9. Coagulation disorder contraindicating intramuscular vaccination.
10. Clinically significant findings on review of systems (determined by investigator or sub-investigator to be sufficient for exclusion).
11. Developmental delay or neurological disorder.
12. Any condition which, in the opinion of the investigator, would interfere with the evaluation of the vaccine or pose a health risk to the subject.
13. History of Hib, diphtheria, tetanus, pertussis or poliovirus disease.

Ages: 42 Days to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 253 (Actual)
Dates: Start 2010-05; Primary Completion 2010-07 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Descriptive statistics will be used to summarize the safety and immunogenicity of the two mixed primary immunization schedules. | serology at 2 and 7 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Langley, MD, Principal Investigator — Dalhousie University
Locations (2):
- Canada (2):
  - Canadian Center for Vaccinology, Halifax, Nova Scotia
  - MUHC- Vaccine Study Centre, Pierrefonds, Quebec

REFERENCES:
- [Derived] Langley JM, Halperin SA, Rubin E, White C, McNeil S, Mutch J, Mackinnon-Cameron D, Smith B. Safety and immunogenicity of 2 mixed primary infant immunization schedules of pentavalent diphtheria, tetanus, acellular pertussis, inactivated poliomyelitis, and Haemophilus influenzae Type B vaccines at 2, 4, and 6 months of age: a randomized controlled trial. Pediatr Infect Dis J. 2012 Feb;31(2):189-92. doi: 10.1097/INF.0b013e318242462a. PMID 22173143